CLINICAL TRIAL: NCT03683927
Title: The Impact of Probiotics in the Respiratory and Gastrointestinal Microbiome and Its Role in Respiratory Tract Infections in Children
Brief Title: Probiotics, Respiratory and Intestinal Microbiome and Respiratory Tract Infections in Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Rosa Maria Wong Chew, Professor B. Head of the Infectious Diseases Research Laboratory, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CONACYT PN 2015-01-878
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Infections in Children
Keywords: Respiratory infections; Probiotics; Microbiome; Viruses; Children
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases | interventions — clausin peptide, Bacillus clausii

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Probiotics consist on Bacillus clausii in a plastic vial that will be administered to the infant 4 times a week
  Interventions: Combination Product: Bacillus clausii
- Placebo group (Placebo Comparator): Sterile water contained in a plastic vial will be administered to the infant 4 times a week
  Interventions: Other: Sterile water

INTERVENTIONS:
Combination Product: Bacillus clausii — The probiotic (Bacillus clausii) will be administered 4 times a week to the infant
  Arms: Probiotics
Other: Sterile water — The placebo group will receive sterile water 4 times a week
  Arms: Placebo group

SUMMARY:
Pneumonia and diarrhea are the most frequent causes of infectious diseases in children under 5 years of age worldwide, responsible for 1.5 million deaths annually.

In up to 80% of pneumonia cases the etiology is viral. Some viruses can persist up to 6 months after an acute infection. The time when viruses enter the body and whether they are commensals or only cause disease and are eliminated after an acute infection is unknown.

Modern techniques have identified diverse communities of microbiota in healthy and sick people, and viral communities associated in a close interaction. The acquisition and colonization by respiratory viruses and the role in health and disease in this niche that is the microbiome is unknown.

The role of probiotics in the prevention of respiratory disease and in the maintenance of homeostasis in the microbiota is poorly understood, and even more the probable relationship between the microbiota, the respiratory viruses that could be commensals or pathogens at the respiratory level, the time when children can be colonized, and their regulation with the administration of probiotics.

The aims of the study are to determine the changes in the intestinal and respiratory microbiota, the viruses that can be commensals or cause disease and the role of probiotics in the prevention of respiratory diseases during the first year of life.

A prospective, randomized, controlled clinical trial will be carried out making basic metagenomics studies (translational medicine). After informed consent, 120 newborns will be randomized into 2 groups, one will receive probiotics 4 times a week orally and the other a placebo consisting of sterile water 4 times a week. The clinical follow up will be done every 2 months until 1 year old, nasal washes and stool samples will be collected to determine the intestinal and respiratory microbiome. Multiplex polymerase chain reaction studies will be conducted to detect the presence of respiratory viruses and the time when the children acquire viruses that are commensal or only in the case of respiratory infection. The mothers will be asked to come for consult in case of respiratory infection and a nasal wash and stool sample will be taken. Descriptive, bivariate and multivariate statistics will be used to determine the associations between the microbiota, the viral metagenomics, the respiratory viruses and the risk of presenting or not respiratory infection in the group receiving probiotics compared to placebo.

DETAILED DESCRIPTION:
Pneumonia and diarrhea are the 2 most frequent causes of infectious diseases in children under 5 years of age worldwide, responsible for 1.5 million deaths annually. In 2013, they corresponded to 15% and 9%, respectively, of the 6.3 million deaths in children under 5 years of age. In our country according to the Ministry of Health, acute respiratory infections are the leading cause of disease nationwide with 27,493, 239 cases reported in 2014 in which pneumonia ranks 19th in the top 20 causes of disease with 174,748 cases, of which 51,893 cases (29%) are in children under 5 years of age, and 21,404 cases (12%) in children under 1 year old; in 2015, 148,140 cases of pneumonia were reported.

It is estimated that in up to 80% of pneumonia cases the etiology is viral. It has been reported that some viruses such as adenovirus or bocavirus can persist up to 6 months after an acute infection. The time when viruses enter the body and whether they are commensals of the respiratory tract or only cause disease and are eliminated after an acute infection is unknown.

Modern techniques have identified diverse communities of microbiota in healthy and sick people, and viral communities associated in a close interaction, which has changed concepts of pathogenesis of respiratory tract infections. The interaction of respiratory viruses, the acquisition and colonization by respiratory viruses and the role in health and disease in this niche that is the microbiome is not known.

The role of probiotics in the prevention of respiratory disease and in the maintenance of homeostasis in the microbiota is poorly studied, and even more the probable relationship between the microbiota, the viroma, the respiratory viruses that could be commensals or pathogens at the respiratory level, the time when children can be colonized, and their regulation with the administration of probiotics.

The aims of the study are to determine the changes in the intestinal and respiratory microbiota, the intestinal and respiratory viroma, the viruses that can be commensals or cause disease and the role of probiotics in the prevention of respiratory diseases during the first year of life.

Methods A prospective, randomized, controlled clinical trial will be carried out making basic metagenomics studies applied to the clinic (translational medicine). In this study the investigators plan to follow up a cohort of 120 children from newborns to one year of age. After informed consent, children will be randomized into 2 groups, one will receive probiotics 4 times a week orally and the other a placebo consisting of sterile water 4 times a week. The clinical follow up will be done every 2 months, where nasal washes and stool samples will be collected to determine the intestinal and respiratory microbiome and the viral metagenomics. Multiplex polymerase chain reaction studies will be conducted to detect the presence of respiratory viruses and detect the time when the children acquire viruses that are commensal or only in case of respiratory infection with manifestations of disease. The mothers will document and will be asked to come for consult in case of respiratory infection, in which samples of nasal washes will be taken to determine the virus or bacteria that could be causing the infection. Descriptive, bivariate and multivariate statistics will be used to determine the associations between the microbiota, the viral metagenomics, the respiratory viruses and the risk of presenting or not respiratory infection in the group receiving probiotics compared to placebo. A p< 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Heathy term newborns
* Vaginal or cesarean section delivery
* Informed consent of both parents to participate

Exclusion Criteria:

* Preterm newborns
* Co-morbidities

Ages: 3 Hours to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-01-09 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Number of respiratory infections in the first year of life | 1 year
  Follow up of the infants will be performed every 2 months during 1 year to look at the incidence of respiratory tract infections in each arm

SECONDARY OUTCOMES:
Rates of bacterial phyla in nasal and intestinal washes | 1 year
  Nasal washes and stool samples will be taken and analyzed for the microbiome. The proportion of phyla will be compared between the probiotic and placebo groups.
Number of viruses detected in nasal washes during the follow up | 1 year
  Nasal washes will be taken every 2 months during 1 year to detect by multiplex polymerase chain reaction viruses that could be in the nasopharynx of the children

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Wong-Chew, MD, DSc, Principal Investigator — Facultad de Medicina, Universidad Nacional Autonoma de Mexico
Locations (1):
- Rosa Maria Wong-Chew, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No